CLINICAL TRIAL: NCT02860702
Title: A Randomized Controlled Trial to Evaluate Growth Velocity and Clinical Outcomes of Infants With Single Ventricle Physiology Fed an Exclusive Human Milk Diet With Early Nutritional Fortification Following Surgical Repair
Brief Title: Exclusive Human Milk Feeding in Infants With Single Ventricle Physiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Prolacta Bioscience (Industry); Baylor College of Medicine (Other); Children's Hospital Medical Center, Cincinnati (Other); Columbia University (Other); University of Oklahoma (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Cook Children's Medical Center (Other); Children's Hospital of Orange County (Other); University of Texas (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC20150779H
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Congenital Heart Defect
Keywords: Single Ventricle; Congenital Heart Defect
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exclusive Human Milk (Experimental): All infants randomized to this arm will receive exclusive human milk diet with addition of human milk derived fortifier from birth to 30 days post initiation of feedings after initial palliative cardiac surgery
  Interventions: Other: Human Milk Derived Fortifier
- Human/Bovine Milk (Active Comparator): All infants randomized to this arm will receive exclusive human milk diet prior to randomization and will use either human and/or bovine milk and fortifier per the institution's standard practice 30 days post initiation of feedings after initial palliative cardiac surgery
  Interventions: Other: Human/Bovine Milk

INTERVENTIONS:
Other: Human Milk Derived Fortifier — Human milk derived fortifier will be utilized to increase caloric intake in infants assigned to the exclusive human milk arm
  Arms: Exclusive Human Milk
Other: Human/Bovine Milk — Bovine milk derived fortification
  Other Names: Human/Formula Milk
  Arms: Human/Bovine Milk

SUMMARY:
A randomized, blinded, controlled trial to evaluate growth velocity and clinical outcomes in infants with single ventricle physiology fed an exclusive human milk diet prior to, and throughout the post-operative period following, surgical repair. Human milk is defined as expressed human milk or donor milk and its derivatives, human milk-based fortifier and human milk caloric fortifier.

The study hypothesis is that infants fed an exclusive human milk diet will have short and long term benefits, with improved wound healing, growth, and neurodevelopmental outcomes while reducing episodes of feeding intolerance and necrotizing enterocolitis (NEC).

DETAILED DESCRIPTION:
This is a single blinded (physician investigator), randomized, controlled trial to evaluate growth velocity and clinical outcomes in infants with single ventricle physiology fed an exclusive human milk diet during their initial hospitalization after birth and through the 30 days post-surgical repair feeding period or hospital discharge, whichever comes first.

Subjects will be randomized to one of two groups at birth or immediately following diagnosis if prenatal care was not obtained prior to birth. Parents who decline participation by their infants in the study will be asked to consent to data gathering on their infants who will be treated and fed per institutional practice. The data on these individuals will be summarized and evaluated descriptively in comparison with the actual trial results.

All patients will receive exclusive maternal human milk or donor human milk prior to randomization. Once randomized, patients in Group One will receive an exclusive human milk diet prior to the surgery and throughout the 30-day feeding period following surgical repair or until hospital discharge, whichever comes first. Day 1 is defined as the day of the first enteral feed post-surgery. Patients in Group Two (Control Group) will receive maternal human milk or formula or donor human milk (per standard of care at each hospital) in the pre-surgical period. In the post-surgical period the control group will receive human milk or formula, as per feeding algorithm The primary objective of this study is to evaluate growth velocity (weight velocity [g/kg/day] and weight z-score from World Health Organization (WHO) growth charts) at 30 days after the initiation of feed post-surgery for infants with single ventricle physiology who are fed an exclusive human milk diet from birth through the 30 day feeding period following surgical repair or until hospital discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Term infants (≥37 and 0/7 weeks gestational age) ≤ 7 days old with a diagnosis of single ventricle physiology who are thought to require a single ventricle repair at the time of enrollment.
2. Infant feeding was NPO or consisted of 100% human milk diet prior to enrollment
3. Parent(s) willing to sign informed consent.
4. Parent(s) willing to comply with study follow-up procedures.
5. Require surgical palliation within the first 1 month of life.

Exclusion Criteria:

1. Term infants >7 days old at the time of diagnosis.
2. <37 weeks gestation
3. Infants requiring cardio-pulmonary resuscitation prior to surgical repair.
4. Outborn infants who received enteral nutrition at the other institution prior to surgical repair. If it is uncertain if infant received even 1 bottle or a small amount of formula, infants will be excluded.
5. Major congenital abnormalities that could significantly affect survival such as:

   1. Confirmed or suspected major genetic abnormalities (lethal or with extremely low probability for survival).
   2. Chromosomal abnormalities: Trisomies (13, 18, 21 etc.) deletions or translocations (Turner/Williams Syndrome, DiGeorge, to name a few)
   3. Major organ system abnormalities not related to a genetic syndrome that are lethal or have extremely low probability for survival (i.e, bilateral kidney intrinsic disease, pulmonary hypoplasia, Central Nervous System (CNS) malformations: Arnold Chiari, myelomeningoceles, hydranencephaly, schizencephaly, holoprosencephaly))
   4. Heterotaxia
   5. Metabolic disorders affecting growth: homocystinuria, methylmalonic acidemias, propionic acidemias, urea cycle defects
6. Evidence of intracerebral hemorrhage (IVH) ≥ Grade 3
7. Any comorbidity or significant clinical event prior to enrollment, deemed by the Investigator as likely to affect survival.
8. Requires Extracorporeal Membrane Oxygenation (ECMO) pre-operatively
9. Legally Authorized Representative(s) unwilling to comply with an exclusive human milk diet either in the form of mother's milk, human milk-based human milk fortifier, human milk based caloric fortifier or donor human milk during the initial hospitalization period and through the 30 day feeding period after surgical repair or hospital discharge, whichever comes first.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
growth velocity | 30 days
  weight velocity in g/kg/day
growth velocity | 30 days
  weight z-score 30 days post 1st operation

SECONDARY OUTCOMES:
linear growth rate | 6 months
  cm/week
linear growth rate | 6 months
  z-score
head circumference growth rate | 6 months
  cm/week
head circumference growth rate | 6 months
  z-score
Feeding Intolerance | 30 days
  defined as nil per os (NPO) for at least 24 in the 30 days of post-surgery enteral feeding period (day 1 is the first day of feeding post-op), NPO due to elective surgeries or procedures will not be defined as feeding intolerance.
Length of stay | up to 24 months
  time hospitalized after 1st surgery
Sepsis | 30 days
  Sepsis 30 days post 1st operation
Necrotizing enterocolitis | 30 days
  NEC 30 days post 1st operation
wound infections | 30 days
  wound infection 30 days post 1st operation
wound dehiscence | 30 days
  wound dehiscence 30 days post 1st operation
parenteral nutrition | 30 days
  in days, during the 30 day post 1st operation

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Blanco, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (12):
- United States (12):
  - Loma Linda University, Loma Linda, California
  - Los Angeles Children's Hospital, Los Angeles, California
  - Children's Hospital Orange County, Orange, California
  - University of Florida Children's Hospital, Gainesville, Florida
  - Lurie Children's Hospital, Chicago, Illinois
  - Columbia University, New York, New York
  - Cincinatti Children's Hospital Medical Center, Cincinnati, Ohio
  - OU Children's Hospital at OU Medical Center, Oklahoma City, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University Health System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
It is a blinded study

REFERENCES:
- [Derived] Blanco CL, Hair A, Justice LB, Roddy D, Bonagurio K, Williams PK, Machado D, Marino BS, Chi A, Takao C, Gordon EE, Ashrafi A, Cacho N, Pruetz JD, Costello JM, Cooper DS; Cardiac Neonate Nutrition Study Group. A Randomized Trial of an Exclusive Human Milk Diet in Neonates with Single Ventricle Physiology. J Pediatr. 2023 May;256:105-112.e4. doi: 10.1016/j.jpeds.2022.11.043. Epub 2022 Dec 14. PMID 36528055